CLINICAL TRIAL: NCT04373811
Title: Quality of Life and Functional Prognosis at One Year of Patients With COVID-19 Admitted in Post-ICU Setting
Brief Title: One-Year Quality of Life and Functional Prognosis of COVID-19 Patients in Post-ICU Setting
Acronym: COVENTRY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Hopital Forcilles (Other)
Responsible Party: Sponsor
Other Study IDs: COVENTRY
Record Dates: First submitted 2020-04-26; First posted 2020-05-04 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; ICU Acquired Weakness; Weaning Failure
Keywords: COVID-19; ICU; ICUAW; Lung Ultrasound; Muscle Ultrasound; Quality of life; Physiotherapy; Diaphragm Ultrasound
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Principal cohort: Quality of life, autonomy and survival will be assessed at one year on 50 patients.
  Safety of early mobilization in post-ICU setting and Medical Reasearch Council (MRC) sum score will be assessed during hospitalization.
- Lung cohort: Lung Ultrasound will be carried out on the first 38 patients of the principal cohort.
  Interventions: Diagnostic Test: Lung ultrasound
- Muscle cohort: Muscle Ultrasound will be carried out on the first 27 patients of the principal cohort.
  Interventions: Diagnostic Test: Muscle ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound will be performed in 12 thorax area: anterior, lateral and posterior, each area divided in superior and inferior area, for each hemithorax.
  Lung Ultrasound Score (lung aeration) will be recorded using a convex probe with a transverse view. Presence of pleural thickening and subpleural consolidations will be recorded.
  Groups: Lung cohort
Diagnostic Test: Muscle ultrasound — Diaphragm ultrasound will be performed using intercostal view with a linear probe at the zone of apposition for assessing diaphragm thickness and thickening and subcostal anterior view with convex probe to assess diaphragm excursion.
  Thickness of vastus intermedius, rectus femori and tibialis anterior will be measured using ultrasound linear probe. Cross-sectionnal area and echogeneicity of rectus femori and tibialis anterior will be measured using ultrasound linear probe. Penation angle of rectus femori will be assessed using ultrasound linear probe.
  Groups: Muscle cohort

SUMMARY:
The COVID-19 disease has been subject to numerous publications since its emergence. Almost 20% of people suffering from COVID-19 develop severe to critical symptoms and require hospitalization, often in Intensive Care Unit (ICU). Respiratory failure is the main reason for admission in ICU of these patients. Therapeutic strategies implemented for the management of critically-ill patients may often lead to short-term muscular and functional alterations resulting in ICU-Acquired Weakness (ICUAW). These lead to long-term disabilities expressing trough dependence and quality of life impairment of survivors.

The purpose of this study is to assess the quality of life, dependence and survival at one year in patients who survived from COVID-19 in ICU and are admitted in post-ICU setting for difficult weaning purpose.

Ancillary studies aim to assess the course of muscle function (atrophy, structural modifications), lung function (loss of aeration) and safety of early mobilization.

DETAILED DESCRIPTION:
SARS-Cov-2, a virus causing a new infectious disease called COVID-19, has been subject to numerous publications since its emergence. Almost 20% of people infected with SARS-Cov-2 develop severe to critical symptoms and required hospitalization, often in Intensive Care Unit (ICU).

Respiratory failure is the main reason for admission in ICU of patients with COVID-19, which develop an Acute Respiratory Distress Syndrome (ARDS). Respiratory failure may be associated to liver, renal, coagulation and hemodynamic failure.

Therapeutic strategies implemented for the management of critically-ill patients with COVID-19 may often lead to short-term muscular and functional alterations resulting in ICU-Acquired Weakness (ICUAW), as studied in other ICU population.

The muscular and functional impairments of patients are associated to a longer duration of mechanical ventilation and hospital length of stay and increased mortality. Long-term impacts are also reported like dependence and quality of life impairment of survivors.

The COVID-19 pandemic currently leads to an increasing number of ICU admission in France with a high risk of settings saturation. Specialized settings for post-ICU rehabilitation are preparing to early receive difficult-to-wean patients with ICUAW after admission in ICU for severe or critical form of COVID-19.

To our best knowledge, no data is obviously available regarding at the future of these patients in terms of quality of life, dependence or survival. Moreover, no short-term data are available concerning the course of lung damages and muscle function after ICU stay. The safety of early mobilization usually delivered in patients admitted to post-ICU settings has never been assessed in patients with COVID-19.

The purpose of this study is to assess the quality of life, dependence and survival at one year in patients who survived from COVID-19 in ICU and are admitted in post-ICU setting for difficult weaning purpose.

Ancillary studies aim to assess course of muscle function (atrophy, structure modification), lung function (loss of aeration) and safety of early mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Patient initially hospitalized in ICU for COVID-19;
* Admitted in post-ICU setting (difficult-to-wean unit);
* Age > 18 years old;
* Membership of a social insurance sheme;
* Medical prescription of early mobilization;
* Patient or relative provides consent.

Exclusion Criteria:

* Known pregnancy ;
* Person subject to judicial health protection;
* Patient under legal guardianship or curatorship;
* Contraidication for early mobilization;
* Decision to withhold lifesustaining treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were initially hospitalized in ICU for COVID-19 and then admitted in a post-ICU setting for difficult weaning purpose.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean in quality of life score at one year on the Short Form Health Survey (SF-36) | 1 year
  Quality of life will be assessed using Short Form Health Survey (SF-36) through a phone call at one year. SF-36 score range from 0 to 100, 100 indicating a better quality of life.

SECONDARY OUTCOMES:
Mean in autonomy score on the Activities Daily Living (ADL) scale | At enrollement and 1 year
  Autonomy will be assessed using Activities Daily Living (ADL) scale through a phone call at one year and six months.
  ADL scale range from 0 to 6, 6 indicating a better autonomy in activities daily living.
Survival rate | 1 year
  Survival will be assessed using the death registry query and phone call for vital status recording at six months and one year. Survival rate will be expressed as a survival function using Kaplan Meier method.
Change from baseline in lung ultrasound aeration score | Day of enrollement, day 14, day 21, day 28 and day 35 from initial admission in ICU
  Lung aeration will be assessed using the Lung Ultrasound Score (LUS). Patient is in semi-recumbent position (30°). Lung ultrasound will be performed in 12 thorax area: anterior, lateral and posterior, each area divided in superior and inferior area, for each hemithorax.
  Lung Ultrasound Score will be recorded using a convex probe with a transverse view.
  For each thorax area a subscore is calculated: 0 = normal profil; 1 = multiple and well-defined B-lines; 2 = confluent B-lines; 3 = lung consolidation.
  Sum of this subscores allows calculation of the total score out of 60. Presence of pleural thickening and subpleural consolidations will be also recorded.
Change from baseline in diaphragm ultrasound thickness and excursion | Day of enrollement, day 14, day 21, day 28 and day 35 from initial admission in ICU
  Diaphragm Ultrasound will be used to assess diaphragm thickness and excursion. Patient is in semi-recumbent position (30°). Diaphragm thickness will be performed using intercostal view with a linear probe at the zone of apposition for assessing diaphragm thickness. M-Mode will be used to measure diaphragm thickness at inspiratory time (maximal inspiration) and expiratory time (maximal expiration).
  Diaphragm excursion will be measured using a subcostal anterior view with convex probe. Excursion measurement is performed in M-mode as the distance between end-inspiration and end-expiration.
  Three measures of both DTF and excursion will performed and the better will be kept.
Mean change from baseline in ultrasound muscle thickness | Day of enrollement, day 14, day 21, day 28 and day 35 from initial admission in ICU
  Muscle ultrasound measurements will be performed using a linear probe with a transverse view.
  Thickness (cm) of vastus intermedius, rectus femori and tibialis anterior will be measured.
Mean change from baseline in ultrasound muscle cross-sectionnal area | Day of enrollement, day 14, day 21, day 28 and day 35 from initial admission in ICU
  Muscle ultrasound measurements will be performed using a linear probe with a transverse view.
  Cross-sectionnal area (CSA) (cm^2) of rectus femori and tibialis anterior will be measured.
Mean change from baseline in ultrasound muscle echogeneicity | Day of enrollement, day 14, day 21, day 28 and day 35 from initial admission in ICU
  Muscle ultrasound measurements will be performed using a linear probe with a transverse view.
  Echogeneicity (0 to 255) of rectus femori and tibialis anterior will be measured using Image J software. Penation angle of rectus femori will be assessed.
  is used to measure muscle thicknesses, CSA and echogeneicity. Longitudinal view is used to measure angle of pennation.
Mean change from baseline in ultrasound muscle pennation | Day of enrollement, day 14, day 21, day 28 and day 35 from initial admission in ICU
  Muscle ultrasound measurements will be performed using a linear probe with a longitudinal view.
  Penation angle (°) of rectus femori will be assessed.
Mean change from baseline in Medical Research Council (MRC) sum score | Day of enrollement, day 14, day 21, day 28 and day 35 from initial admission in ICU
  MRC sum score evaluates strength in three muscle groups of all four limbs. A score between 0 and 5 is assigned to each of them, which renders a maximum total score of 60.
Prevalence of adverse outcomes during early mobilization | From date of enrollement up to 30 days (date of estimated post-ICU discharge)
  Number of adverse outcomes during early mobilization of patients will recorded at each mobilization session. Prevalence of adverse outcomes is expressed as the number of adverse outcomes divided by the number of early mobilization sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric LE NEINDRE, PT, PhD, Principal Investigator — Hopital Forcilles
Locations (3):
- France (3):
  - Centre Hospitalier de Béthune, Beuvry, Hauts-de-France
  - Hôpital Forcilles, Férolles-Attilly, Île-de-France Region
  - APHP - Hôpital Universitaire Pitié-Salpétrière, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be openly available in "figshare".
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at publication of the results.
Access Criteria: Data openly available in a public repository that issues datasets with DOIs

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Murthy S, Gomersall CD, Fowler RA. Care for Critically Ill Patients With COVID-19. JAMA. 2020 Apr 21;323(15):1499-1500. doi: 10.1001/jama.2020.3633. No abstract available. PMID 32159735
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Herridge MS, Moss M, Hough CL, Hopkins RO, Rice TW, Bienvenu OJ, Azoulay E. Recovery and outcomes after the acute respiratory distress syndrome (ARDS) in patients and their family caregivers. Intensive Care Med. 2016 May;42(5):725-738. doi: 10.1007/s00134-016-4321-8. Epub 2016 Mar 30. PMID 27025938
- [Background] Bouhemad B, Liu ZH, Arbelot C, Zhang M, Ferarri F, Le-Guen M, Girard M, Lu Q, Rouby JJ. Ultrasound assessment of antibiotic-induced pulmonary reaeration in ventilator-associated pneumonia. Crit Care Med. 2010 Jan;38(1):84-92. doi: 10.1097/CCM.0b013e3181b08cdb. PMID 19633538
- [Background] Peng QY, Wang XT, Zhang LN; Chinese Critical Care Ultrasound Study Group (CCUSG). Findings of lung ultrasonography of novel corona virus pneumonia during the 2019-2020 epidemic. Intensive Care Med. 2020 May;46(5):849-850. doi: 10.1007/s00134-020-05996-6. Epub 2020 Mar 12. No abstract available. PMID 32166346
- [Background] Parry SM, El-Ansary D, Cartwright MS, Sarwal A, Berney S, Koopman R, Annoni R, Puthucheary Z, Gordon IR, Morris PE, Denehy L. Ultrasonography in the intensive care setting can be used to detect changes in the quality and quantity of muscle and is related to muscle strength and function. J Crit Care. 2015 Oct;30(5):1151.e9-14. doi: 10.1016/j.jcrc.2015.05.024. Epub 2015 Jun 3. PMID 26211979
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Flaatten H, Kvale R. Survival and quality of life 12 years after ICU. A comparison with the general Norwegian population. Intensive Care Med. 2001 Jun;27(6):1005-11. doi: 10.1007/s001340100960. PMID 11497132
- [Background] Cartwright MS, Kwayisi G, Griffin LP, Sarwal A, Walker FO, Harris JM, Berry MJ, Chahal PS, Morris PE. Quantitative neuromuscular ultrasound in the intensive care unit. Muscle Nerve. 2013 Feb;47(2):255-9. doi: 10.1002/mus.23525. Epub 2012 Oct 5. PMID 23041986